CLINICAL TRIAL: NCT03820414
Title: A Phase 1, Randomized, Placebo-Controlled, Observer-Blind, Antigen Dose-Escalation and Adjuvant Dose-Ranging Clinical Trial to Evaluate the Safety, Tolerability, and Immunogenicity of CRV-101 in Healthy Adult Subjects
Brief Title: Safety, Tolerability, and Immunogenicity of CRV-101 in Healthy Adult Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Curevo Inc (Industry)
Collaborators: Access to Advanced Health Institute (AAHI) (Other); Mogam Biotechnology Research Institute (Unknown); Green Cross Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CRV-101-100
Record Dates: First submitted 2019-01-24; First posted 2019-01-29 (Actual); Last update posted 2021-02-11 (Actual); Status verified 2021-02

CONDITIONS: Herpes Zoster; Varicella Zoster
Keywords: VZV, Vaccine, Shingles
MeSH Terms: conditions — Herpes Zoster | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- CRV101 Group 1 (Experimental): Subjects receive 2 doses of the candidate CRV-101 formulation 1, administered intramuscularly (IM) in deltoid region of non-dominant arm, according to a 0, 2 Month schedule.
  Interventions: Biological: CRV 101
- CRV 101 Group 2 (Experimental): Subjects receive 2 doses of the candidate CRV-101 formulation 2, administered intramuscularly (IM) in deltoid region of non-dominant arm, according to a 0, 2 Month schedule.
  Interventions: Biological: CRV 101
- CRV 101 Group 3 (Experimental): Subjects receive 2 doses of the candidate CRV-101 formulation 3, administered intramuscularly (IM) in deltoid region of non-dominant arm, according to a 0, 2 Month schedule.
  Interventions: Biological: CRV 101
- CRV 101 Group 4 (Experimental): Subjects receive 2 doses of the candidate CRV-101 formulation 4, administered intramuscularly (IM) in deltoid region of non-dominant arm, according to a 0, 2 Month schedule.
  Interventions: Biological: CRV 101
- Control Group (Placebo Comparator): Subjects received 2 doses of placebo (saline solution), administered intramuscularly (IM) in deltoid region of non-dominant arm, according to a 0, 2 Month schedule.
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: CRV 101 — (Different formulations)
  Arms: CRV 101 Group 2; CRV 101 Group 3; CRV 101 Group 4; CRV101 Group 1
Biological: Placebo — 2 doses administered IM in deltoid region of non-dominant arm
  Other Names: Saline injection
  Arms: Control Group

SUMMARY:
The purpose of this clinical trial is to evaluate the safety, tolerability, and immunogenicity of vaccine candidate CRV-101, investigational vaccine in healthy adult subjects in the United States.

ELIGIBILITY:
Inclusion Criteria:

1. Males and non-pregnant females ≥ 18 to < 50 years of age at the time of enrollment.
2. In good general health as confirmed by a medical history and physical exam, vital signs*, and screening laboratories conducted no more than 30 days prior to study injection administration.

   *Oral Temperature <38°C, respiratory rate < 17 breaths pm, heart rate ≤100 bpm and >54 bpm, systolic blood pressure ≤150 mmHg and >89 mmHg, diastolic blood pressure ≤95 mmHg.

   NOTE: Athletically trained subjects with a heart rate ≥40 may be enrolled at the discretion of the principal investigator or designated licensed clinical investigator and reasoning must be documented.
3. Screening laboratory values must be within normal range or not clinically significant as determined by the PI and approved by the Medical Monitor: sodium, potassium, BUN, ALT, AST, total bilirubin, alkaline phosphatase, creatinine, random glucose, WBC with differential, hemoglobin, and platelet count.
4. Negative HIV 1/2 antibody, hepatitis B surface antigen (HBsAg), and hepatitis C virus (HCV) antibody.
5. Normal urinalysis or if abnormal determined to be not clinically significant by the PI and the Medical Monitor (trace protein is acceptable without medical monitor approval).
6. Urine test result for recreational drugs/drugs of abuse that in the opinion of the PI would not be a concern for subject's safety, or ability to reliably attend visits, and perform required protocol procedures. If urine drug test is positive, reasoning for inclusion must be documented.
7. Females of childbearing potential* must have a negative serum pregnancy test at screening and a negative urine pregnancy test on the day of each study vaccination (prior to vaccination), must not be breast-feeding, and women in sexual relationships with men must agree to practice acceptable contraception** for the 30-day period before Day 0 through 90 days after the last study injection. These precautions are necessary due to unknown effects that CRV-101 might cause in a fetus or newborn infant.

   *Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or < 1 year of the last menses if menopausal). Post-menopausal defined as at least 12 months spontaneous amenorrhea and confirmed with FSH > 40 mIU/ml.

   **Includes, but is not limited to, sexual abstinence, monogamous relationship with vasectomized partner who has been vasectomized for 6 months or more prior to the subject receiving study product, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing ®, and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill").
8. Exposure to VZV as documented by one of the following: subject reported clinical history of chickenpox, previous vaccination against VZV with Varivax® (or other low-titer live-attenuated varicella vaccine), or positive serology test for VZV.
9. Must be able to understand informed consent in English and capable of completing a study diary card in English.
10. Must provide informed consent prior to any screening procedures performed, be able and willing to make all study visits, be reachable by telephone or personal contact by the study site personnel, and have a permanent address.
11. Willing to abstain from donating whole blood or blood derivatives until after Day 365 visit.

Exclusion Criteria:

1. History of chickenpox or herpes zoster in the past 3 years.
2. Immunization with a vaccine against herpes zoster (Zostavax® or Shingrix®).
3. Participation in another experimental protocol with last receipt of any device, vaccine, or other immunomodulator investigational products within the past 180 days of enrollment, or last receipt of non-device, non-vaccine, non-immunomodulator investigational products with in the last 90 days of enrollment or 5 half-lives whichever is greater, or planned participation in any other investigational study during the study period.
4. Chronic administration (defined as more than 14 days in total) of immunosuppressants or other immune-modifying drugs (e.g. oral or injected steroids, such as prednisone; high dose inhaled steroids; biologics (e.g. TNF inhibitor, or other cytokine inhibitors) or cytotoxic therapies, such as chemotherapy drugs or radiation) within 180 days prior to enrollment and during the study through Day 365 visit. For corticosteroids, this will mean prednisone ≥ 0.5 mg/kg/day, or equivalent. Low dose inhaled and topical steroids are allowed.
5. Received a blood transfusion or immunoglobulin within past 90 days of enrollment.
6. Donated blood products (platelets, whole blood, plasma, etc.) within past 60 days of enrollment.
7. Received any vaccine within past 30 days prior to enrollment and no planned immunizations while on study with the exception of seasonal influenza vaccine which must not be given until 30 days after the last study injection and the Day 84 immunology blood has been drawn and a 30 day window prior to each immunology blood draw (Day 196, 365).
8. History of autoimmune disease or other causes of immunosuppressive states.
9. History of any acute or chronic illness (including cardiovascular, pulmonary, neurological, hepatic, rheumatic, hematological, metabolic or renal disorders, controlled hypertension), or use of medication that, in the opinion of the Principal Investigator, may interfere with the evaluation of the safety or immunogenicity of the vaccine.
10. Rash, tattoos, or any other dermatological condition that could adversely affect the vaccine injection site or interfere with its evaluation.
11. BMI that poses a health risk in the opinion of the Principal Investigator.
12. Hypertension (systolic >150 or diastolic >95).
13. History of significant psychiatric illness (including past history of suicidal ideation or attempt) with or without current use of medication.
14. Known or suspected alcohol or drug abuse within the past 5 years.
15. Chronic smoker (> 20 pack years).
16. Subjects with a history of previous anaphylaxis or severe allergic reaction to vaccines or unknown allergens.
17. Subjects who are unlikely to cooperate with the requirements of the study protocol or who are likely to be unreliable in attending study visits or other reason that the Principal Investigator determines that the subject will not be a good candidate to participate in this study.

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2019-01-03 (Actual); Primary Completion 2020-04-04 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
The number of subjects experiencing solicited local injection site reactions within 7 days following each study injection. | 7 Days
The number of subjects experiencing solicited systemic reactions within 7 days following each study injection. | 7 Days
The number of subjects spontaneously reporting unsolicited adverse events from Day 0 through 28 days after the last injection. | 28 Days
The number of medically-attended adverse events considered related to any of the study injections reported at any point during the study period events and potential immune-mediated medical conditions considered related to any of the study injections | 421 Days

SECONDARY OUTCOMES:
The frequencies of vaccine protein-specific T cells elicited by the CRV101 study vaccine at specified time points. | Day 0, 7, 28, 56, 63, 84, 196, and 365
The levels of vaccine protein-specific antibodies elicited by the CRV101 study vaccine at specified time points | Day 0, 7, 28, 56, 63, 84, 196, and 365

CONTACTS AND LOCATIONS:
Overall Officials: John E Ervin, MD, Principal Investigator — The Center for Pharmaceutical Research; Corey Casper, MD, Study Director — Access to Advanced Health Institute (AAHI); Lisa Shelton, Study Chair — Curevo Inc
Locations (1):
- The Center for Pharmaceutical Research, Kansas City, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen JI. Clinical practice: Herpes zoster. N Engl J Med. 2013 Jul 18;369(3):255-63. doi: 10.1056/NEJMcp1302674. PMID 23863052